CLINICAL TRIAL: NCT00601263
Title: Center for Chinese Herbal Therapy for Asthma. Project #2-Clinical Effect of a Chinese Herbal Therapy in Human Asthma-Phase I
Brief Title: Safety Study of Chinese Herbal Therapy to Treat Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xiu-Min Li (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Xiu-Min Li, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P01AT002647 (NIH); P01AT002647 (NIH); GCO 04-0206
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2012-02

CONDITIONS: Asthma
Keywords: Chinese Herbal Therapy; Asthma; Investigational new drug (IND); Complementary and Alternative Medicine
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1a (Active Comparator): Low dose ASHMI (2 caps bid).
  Interventions: Drug: Anti-Asthma Herbal Medical Intervention (ASHMI)
- 1b (Placebo Comparator): Placebo 2 caps bid.
  Interventions: Drug: Anti-Asthma Herbal Medical Intervention (ASHMI)
- 2a (Active Comparator): Medium dose ASHMI (4 caps bid).
  Interventions: Drug: Anti-Asthma Herbal Medical Intervention (ASHMI)
- 2b (Placebo Comparator): Placebo 4 caps bid.
  Interventions: Drug: Anti-Asthma Herbal Medical Intervention (ASHMI)
- 3a (Active Comparator): High dose ASHMI (6 caps bid).
  Interventions: Drug: Anti-Asthma Herbal Medical Intervention (ASHMI)
- 3b (Placebo Comparator): Placebo 6 caps bid.
  Interventions: Drug: Anti-Asthma Herbal Medical Intervention (ASHMI)

INTERVENTIONS:
Drug: Anti-Asthma Herbal Medical Intervention (ASHMI) — We propose to test 3 daily doses in which 2,4, or 6 ASHMI or placebo capsules will be administered orally twice daily (BID) for 7 days.

SUMMARY:
The purpose of this study is to determine the safety of an anti-asthma herbal medicine intervention (ASHMI) in adult asthmatics and to see what effects ASHMI has on certain parts of the immune system.

DETAILED DESCRIPTION:
Asthma is a major public health problem worldwide, particularly in westernized societies and has continued to increase in prevalence over the past two decades. Inhaled corticosteroids have become the first-line treatment for persistent asthma even though significant side effects have been reported. New asthma medications, including leukotriene inhibitors and anti-IgE, have shown only marginal benefits. Patients have increasingly turned to complementary and alternative medicine (CAM) for treatment of their asthma, despite the uncertainty of its benefits due a lack of well-controlled scientific studies.

We have developed a Chinese herbal formula composed of 3 herbs called ASHMI. It has been previously shown in murine studies that ASHMI (a formula containing Ling Zhi, Ku Shen and Gan Cao) has therapeutic effects on the major pathogenic mechanisms of asthma-airway hyperreactivity, pulmonary inflammation, and airway remodeling, as well as a down-regulating of TH2 response. A subsequent study in 91 asthmatic patients in Weifang, China found ASHMI to be a safe and effective alternative to prednisone for treating asthma and exhibited a beneficial effect on TH1 and TH2 balance. Based on these preliminary studies, we hypothesize that ASHMI will be a safe medication in atopic patients with asthma and will lead to identifiable changes in serum immunologic markers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ages 18-40 and otherwise in good health as determined by medical history and physical examination
* History of asthma documented by a physician
* Documentation of allergy to two or more common environmental allergens as evidenced by positive prick skin or RAST testing
* The subject agrees to participate in the study
* Females of childbearing potential must be inactive sexually or take effective birth control measures, as deemed appropriate by the investigator, for the duration of the study.

Exclusion Criteria:

* Acute illness (such as cold, flu, etc.) within one week before the administration of study drug
* Any history of systemic disease that in the investigator's opinion would preclude the subject from participating in this study, including viral hepatitis infection (by patient self-report)
* Abnormal hepatic function
* Abnormal bone marrow function
* Abnormal renal function
* Clinically significant abnormal electrocardiogram
* Current uncontrolled moderate to severe asthma with FEV1 <80% predicted
* Participation in another experimental study within 30 days of this study
* History of alcohol or drug abuse (by self report)
* Pregnant or lactating female subjects. Females of childbearing potential will need a negative serum pregnancy test to be considered for this study
* Current smokers

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Drug safety (absence of severe adverse effects) | 1 week

SECONDARY OUTCOMES:
Clinically significant changes in electrocardiogram | 1 week
Clinically significant changes in blood count | 1 week
Clinically significant changes in serum chemistries | 1 week
Clinically significant changes in renal function | 1 week
Clinically significant changes in liver function | 1 week
Clinically significant changes in urinalysis | 1 week
Allergen-specific IgE levels | 1 week
Total IgA level | 1 week
T-cell cytokine profile | 1 week
Prostaglandin levels | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Juan Wisnivesky, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School Medicine, New York, New York, United States

REFERENCES:
- [Background] Wen MC, Wei CH, Hu ZQ, Srivastava K, Ko J, Xi ST, Mu DZ, Du JB, Li GH, Wallenstein S, Sampson H, Kattan M, Li XM. Efficacy and tolerability of anti-asthma herbal medicine intervention in adult patients with moderate-severe allergic asthma. J Allergy Clin Immunol. 2005 Sep;116(3):517-24. doi: 10.1016/j.jaci.2005.05.029. PMID 16159618